CLINICAL TRIAL: NCT00060437
Title: A Phase II Trial Of Oral Perifosine In Patients With Metastatic Androgen Independent Prostate Cancer
Brief Title: Perifosine in Treating Patients With Metastatic, Androgen-Independent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000301951; NCI-03-C-0157; NCI-5970; NCT00058708 (obsolete NCT alias)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2004-04

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — perifosine

INTERVENTIONS:
Drug: perifosine

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as perifosine use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of perifosine in treating patients who have prostate cancer that no longer responds to androgen ablation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 4-month progression-free survival rate, as measured by prostate-specific antigen and clinical criteria, in patients with metastatic androgen-independent prostate cancer treated with perifosine.
* Determine the side-effect profile of this drug in these patients.
* Determine the pharmacokinetics and pharmacodynamics of this drug in these patients.

OUTLINE:

* Course 1: Patients receive oral perifosine twice on day 1 and once daily on days 2-21.
* All subsequent courses: Patients receive oral perifosine once daily on days 1-21.

In all courses, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 22-46 patients will be accrued for this study within approximately 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate, meeting all of the following criteria:

  * Metastatic
  * Androgen-independent
  * Progressive disease while continuing to receive hormonal ablation (e.g., luteinizing hormone-releasing hormone [LHRH] agonist)
* Progression documented by at least 1 of the following parameters:

  * Two consecutively rising prostate-specific antigen levels, at least 1 week apart, with at least 1 measurement that is 50% above the nadir reached after the last treatment regimen (as long as the last measurement is at least 5 ng/mL)
  * At least 1 new metastatic lesion on technetium Tc 99m bone scintigraphy
  * Progression of soft-tissue metastases as measured by appropriate modalities (i.e., imaging or palpation) and demonstrated by at least 1 of the following:

    * Development of new area of malignant disease (measurable or nonmeasurable)
    * At least a 20% increase in the sum of the longest diameters (LD) of target lesions from the smallest sum of LD recorded since the treatment started or the appearance of 1 or more new lesions
* Patients who have not undergone surgical castration must have a testosterone level less than 50 ng/mL and continue on their LHRH agonist during study treatment
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin less than 1.0 mg/dL or upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN

Renal

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No myocardial infarction within the past 6 months
* No unstable or newly diagnosed angina pectoris
* No New York Heart Association class II-IV congestive heart failure

Ophthalmic

* No pre-existing retinal disease
* No pathologic baseline electrooculogram

Other

* Fertile patients must use effective barrier contraception
* Able to ingest oral medication
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to perifosine (e.g., miltefosine or edelfosine)
* No ongoing or active infection
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No other active malignancies within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of the bladder

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 1 prior chemotherapy regimen
* More than 4 weeks since prior chemotherapy (at least 6 weeks for nitrosoureas or mitomycin)

Endocrine therapy

* See Disease Characteristics
* More than 4 weeks since prior flutamide
* More than 6 weeks since prior bicalutamide or nilutamide

Radiotherapy

* At least 6 weeks since prior bone-seeking radioisotopes
* Recovered from prior radiotherapy

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Other

* Recovered from any acute toxicity related to prior therapy
* More than 3 months since prior UCN-01
* More than 3 months since prior suramin
* No concurrent commercial or other investigational agents or therapies intended to treat the malignancy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin M. Posadas, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Posadas EM, Gulley J, Arlen PM, Trout A, Parnes HL, Wright J, Lee MJ, Chung EJ, Trepel JB, Sparreboom A, Chen C, Jones E, Steinberg SM, Daniels A, Figg WD, Dahut WL. A phase II study of perifosine in androgen independent prostate cancer. Cancer Biol Ther. 2005 Oct;4(10):1133-7. doi: 10.4161/cbt.4.10.2064. Epub 2005 Oct 1. PMID 16138006
- [Result] Posadas EM, Trout A, Senderowicz AM, et al.: A phase II trial of oral perifosine in patients with metastatic androgen-independent prostate cancer (AIPC). [Abstract] SUO/NCI Urologic Oncology Meeting, December 5-6, 2003, Bethesda, MD. A-54, 38, 2003.